CLINICAL TRIAL: NCT00410683
Title: Phase III Study Comparing Post-Operative Conformal Radiotherapy to No Post-Operative Radiotherapy in Patients With Completely Resected Non-Small Cell Lung Cancer and Mediastinal N2 Involvement [Lung ART]
Brief Title: Radiation Therapy in Treating Patients With Non Small Cell Lung Cancer That Has Been Completely Removed by Surgery
Acronym: LUNG ART
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: Intergroupe Francophone de Cancerologie Thoracique (Other); The Christie NHS Foundation Trust (Other); European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000523568; 2006/1202 (Other: CSET number); PROTEGE-01/0601 (Other: UNICANCER); 20671 (Other: European Union); IFCT - 0503 (Other: IFCT); UK11/NW/0075 (Other: The Christie NHS Foundation Trust)
Record Dates: First submitted 2006-12-11; First posted 2006-12-13 (Estimated); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Non-small Cell Lung Cancer
Keywords: stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Watchful Waiting; Chemotherapy, Adjuvant; Radiotherapy, Conformal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radiotherapy (Experimental): Beginning within 4-8 weeks after surgery or 2-6 weeks after chemotherapy, patients undergo adjuvant thoracic conformal radiotherapy once daily, 5 days per week, for 6 weeks.
  Interventions: Other: clinical observation; Procedure: adjuvant therapy; Radiation: 3-dimensional conformal radiation therapy
- No radiotherapy (Active Comparator): Patients do not undergo adjuvant thoracic radiotherapy. After completion of study therapy, patients are followed periodically for up to 10 years.
  Interventions: Other: clinical observation; Procedure: adjuvant therapy

INTERVENTIONS:
Other: clinical observation
Procedure: adjuvant therapy
Radiation: 3-dimensional conformal radiation therapy
  Arms: Radiotherapy

SUMMARY:
RATIONALE: Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. Giving radiation therapy after surgery may kill any tumor cells that remain after surgery. It is not yet known whether giving radiation therapy after surgery is more effective than no radiation therapy in treating patients with non-small cell lung cancer.

PURPOSE: This randomized phase III trial is studying radiation therapy to see how well it works compared to no radiation therapy in treating patients with non-small cell lung cancer that has been completely removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the disease-free survival of patients with completely resected non-small cell lung cancer treated with conformal thoracic radiotherapy vs no radiotherapy.

Secondary

* Determine the toxicity, in particular cardiac and pulmonary toxicity, of these regimens in these patients.
* Compare the local control in patients treated with these regimens.
* Determine patterns of recurrence in patients treated with these regimens.
* Determine the overall survival of patients treated with these regimens.
* Assess second cancers in patients treated with these regimens.
* Assess prognostic factors and predictive factors of treatment effect on disease-free survival and overall survival of patients treated with these regimens.
* Determine the cost per recurrence-free year of life.

OUTLINE: This is a multicenter, randomized study.

Patients are stratified according to participating center, prior chemotherapy (neoadjuvant alone vs adjuvant vs none), number of lymph stations involved (0 vs 1 vs ≥ 2), histology (squamous cell vs other), and use of pretreatment positron emission tomography scans (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Beginning within 4-8 weeks after surgery or 2-6 weeks after chemotherapy, patients undergo adjuvant thoracic conformal radiotherapy once daily, 5 days per week, for 6 weeks.
* Arm II: Patients do not undergo adjuvant thoracic radiotherapy. After completion of study therapy, patients are followed periodically for up to10 years.

PROJECTED ACCRUAL: A total of 700 patients will be accrued for this study.

ELIGIBILITY:
INCLUSION CRITERIA :

1. Histological evidence of non-small cell lung cancer (NSCLC)
2. Complete resection by lobectomy, bilobectomy or pneumonectomy (i.e patients with positive margins) or extra-capsular mediastinal nodal extension breaching the surface of the pathological specimen should not to be included
3. Mediastinal lymph node exploration (lymph node sampling or systematic dissection of lymph nodes at stations 2, 4 and 7 in case of upper/middle right-sided lung cancer; 4, 7, 8 and 9 in case of lower right-sided lung cancer; 5, 6 and 7 in case of upper left -sided lung cancer; 7, 8 and 9 in case of lower left-sided lung cancer is recommended)
4. Pathologically or cytologically documented N2 mediastinal nodal involvement, at the time of surgery if no preoperative chemotherapy or before preoperative chemotherapy, according to the criteria of the joint AJCC and UICC classification, clinical N2 patients without cytological or histological documentation of mediastinal node involvement before preoperative chemotherapy can be included in the study if and only if, they have histologically confirmed N2 disease at the time of surgery
5. Prior chemotherapy is allowed (pre-operative or post-operative adjuvant chemotherapy, or both)
6. Patient aged ≥ 18 years
7. Good Performance status (WHO ≤ 2)
8. Fit enough to receive curative radiotherapy
9. Adequate pulmonary function with post-operative FEV1 after surgery > 1 l or over 35% theoretical value
10. Signed informed consent form

EXCLUSION CRITERIA:

1. Documented metastases, (except for ipsilateral nodule(s) in a different lobe after pneumonectomy or bi-lobectomy)
2. Major pleural or pericardial effusion
3. Synchronous contra-lateral lung cancer
4. Clinical progression during post-operative chemotherapy
5. Previous chest radiotherapy
6. Intention of concomitant chemotherapy during radiotherapy
7. Weight loss in the previous 6 months before surgery ≥ 10 %
8. Evidence of severe or uncontrolled systemic disease as judged by the investigator
9. Recent (< 6 months) severe cardiac disease (arrhythmia, congestive heart failure, infarction, pace-maker) or pulmonary disease
10. Current or past history of neoplasm other than non-small cell lung cancer diagnosed within the last 5 years, except :

    * basal cell carcinoma of the skin
    * in situ carcinoma of the cervix A patient diagnosed for another neoplasm 5 years ago or more, treated and considered as cured may be included in the study if all the other criteria are respected.
11. Pregnancy or breast feeding or inadequate contraceptive measures during treatment
12. Patients who, for family, social, geographic or psychological reasons, cannot be adequately followed up and/or are incapable of undergoing regular controls
13. Patient deprived of freedom or under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2007-02 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | assessed up every 3 and 6 months after randomization, every 6 months for the fist three years and yearly afterward

SECONDARY OUTCOMES:
Acute and late toxicity (with identification of predictive factors of toxicity) | assessed up at 3 and 6 months after randomization and then yearly afterward; And in case of event
Local control | assessed up at 3 and 6 months after randomization and then yearly afterward; And in case of event
Patterns of failure | assessed up at 3 and 6 months after randomization and then yearly afterward; And in case of event
Overall survival (OS) | assessed up In case of death whatever the cause
Second cancers | Assessed up in case of event
Prognostic and predictive factors of treatment effect on DFS and OS | assessed up at the end of the study
Cost per recurrence-free year of life | Assessed up at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Cecile Le Pechoux, MD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Institut Gustave Roussy, Villejuif, Val De Marne, France

REFERENCES:
- [Derived] Predina J, Suliman R, Potter AL, Panda N, Diao K, Lanuti M, Muniappan A, Jeffrey Yang CF. Postoperative radiotherapy with modern techniques does not improve survival for operable stage IIIA-N2 non-small cell lung cancer. J Thorac Cardiovasc Surg. 2023 May;165(5):1696-1709.e4. doi: 10.1016/j.jtcvs.2022.09.062. Epub 2022 Oct 18. PMID 36610886
- [Derived] Le Pechoux C, Pourel N, Barlesi F, Lerouge D, Antoni D, Lamezec B, Nestle U, Boisselier P, Dansin E, Paumier A, Peignaux K, Thillays F, Zalcman G, Madelaine J, Pichon E, Larrouy A, Lavole A, Argo-Leignel D, Derollez M, Faivre-Finn C, Hatton MQ, Riesterer O, Bouvier-Morel E, Dunant A, Edwards JG, Thomas PA, Mercier O, Bardet A. Postoperative radiotherapy versus no postoperative radiotherapy in patients with completely resected non-small-cell lung cancer and proven mediastinal N2 involvement (Lung ART): an open-label, randomised, phase 3 trial. Lancet Oncol. 2022 Jan;23(1):104-114. doi: 10.1016/S1470-2045(21)00606-9. Epub 2021 Dec 15. PMID 34919827